CLINICAL TRIAL: NCT01353781
Title: A Phase I, Open-Label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumour Activity of Ascending Doses of AZD5363 Under Adaptable Dosing Schedules in Japanese Patients With Advanced Solid Malignancies
Brief Title: Open Label Phase 1 Study in Japan for Patient With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3610C00004
Record Dates: First submitted 2011-04-11; First posted 2011-05-16 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Advanced Solid Malignancy; Advanced Solid Tumor
Keywords: Phase 1; advanced solid tumor; AKT; Ascending; Japanese
MeSH Terms: interventions — capivasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD5363 (Experimental): Ascending doses of AZD5363 administered orally to patients to define the maximum tolerated dose (MTD)
  Interventions: Drug: AZD5363

INTERVENTIONS:
Drug: AZD5363 — Patients will be given AZD5363 capsules administered orally as a single dose, and then multiple twice-daily dosing following 3 to 7 days washout.

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics and preliminary anti-tumour activity of ascending doses of AZD5363 under adaptable dosing schedules in Japanese patients with advanced solid malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 20 years
* Histological or cytological confirmation of a solid malignant tumour, excluding lymphoma, that is refractory to standard therapies or for which no standard therapies exist
* At least one lesion (measurable and/or non-measurable) that can be accurately assessed according to RECIST
* World Health Organisation (WHO) performance status 0-1 with no deterioration over the previous 2 weeks and minimum life expectancy of 12 weeks
* Patients should be willing to remain in hospital until the completion of the first cycle including cycle 0, cycle 1, and cycle 2 Day1 (as cycle 1 Day 21)

Exclusion Criteria:

* Clinically significant abnormalities of glucose metabolism as defined by any of the following:
* Diagnosis of diabetes mellitus type I or II (irrespective of management)
* Baseline fasting glucose value of ≥7 mmol/l (126mg/dL)
* Glycosylated haemoglobin (HbA1C) >6.5%
* Spinal cord compression or brain metastases unless asymptomatic, treated and stable and not requiring steroids for at least 4 weeks prior to start of study treatment
* Inadequate bone marrow reserve or organ function
* Any evidence of severe or uncontrolled systemic diseases, including active bleeding diatheses, or active infection
* With the exception of alopecia, any unresolved toxicities from prior therapy greater than CTCAE grade 1 at the time of starting study treatment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2011-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
To investigate the safety and tolerability of AZD5363 to define a Recommended Dose (RD) when given orally | All AEs will be collected throughout the study, from informed consent until 30 days after the end of study treatment. The total duration of this time frame can not be specified, as it depends on the number of treatments the subject may receive
  To investigate the safety and tolerability of AZD5363 to define a Recommended Dose (RD) when given orally, either as a continuous or an intermittent schedule, for further clinical evaluation when given to Japanese patients with advanced solid malignancies

SECONDARY OUTCOMES:
To define the maximum tolerated dose (MTD) if possible or biological effective dose in Japanese patients with advanced solid malignancies. | once 2 or more participants experience a DLT a dose level during the study period (within approx 20 months)
  To define the maximum tolerated dose (MTD) if possible or biological effective dose in Japanese patients with advanced solid malignancies. A dose will be considered non-tolerated and dose escalation will cease if 2 or more of up to 6 evaluable patients experience a DLT at a dose level. Six evaluable patients are required to determine the MTD
To characterise the pharmacokinetics parameters Cmin | PK measurements on Cycle 0 Day 1/2/3 and Cycle 1 Day 1/8/15.
  To characterise the pharmacokinetics parameters Cmin of AZD5363 following a single administration and after multiple dosing when given orally to Japanese patients with advanced solid malignancies
To obtain a preliminary assessment of the anti-tumour activity of AZD5363 by evaluation of tumour response using Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1 in Japanese patients with advanced solid malignancies | Assessed every 3 weeks for initial 2 cycles and every 6 weeks for later cycles for all subjects after start of study treatment until discontinuation of study treatment or withdrawal of consent.
  To obtain a preliminary assessment of the anti-tumour activity of AZD5363 by evaluation of tumour response using Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1 in Japanese patients with advanced solid malignancies.
  The total duration of this time frame can not be specified, as it depends on the number of treatments the subject may receive.
To characterise the pharmacokinetics parameters(Cmax) | PK measurements on Cycle 0 Day 1/2/3 and Cycle 1 Day 1/8/15.
  To characterise the pharmacokinetics parameters Cmax of AZD5363 following a single administration and after multiple dosing when given orally to Japanese patients with advanced solid malignancies
To characterise the pharmacokinetics parameters tmax | PK measurements on Cycle 0 Day 1/2/3 and Cycle 1 Day 1/8/15.
  To characterise the pharmacokinetics parameters tmax of AZD5363 following a single administration and after multiple dosing when given orally to Japanese patients with advanced solid malignancies
To characterise the pharmacokinetics parameters AUC | PK measurements on Cycle 0 Day 1/2/3 and Cycle 1 Day 1/8/15.
  To characterise the pharmacokinetics parameters AUC factor of AZD5363 following a single administration and after multiple dosing when given orally to Japanese patients with advanced solid malignancies
To characterise the pharmacokinetics parameters CL/F | PK measurements on Cycle 0 Day 1/2/3 and Cycle 1 Day 1/8/15.
  To characterise the pharmacokinetics parameters CL/F factor of AZD5363 following a single administration and after multiple dosing when given orally to Japanese patients with advanced solid malignancies
To characterise the pharmacokinetics parameters Vz/F | PK measurements on Cycle 0 Day 1/2/3 and Cycle 1 Day 1/8/15.
  To characterise the pharmacokinetics parameters Vz/F of AZD5363 following a single administration and after multiple dosing when given orally to Japanese patients with advanced solid malignancies

CONTACTS AND LOCATIONS:
Overall Officials: Paul Stockman, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, Chūōku, Japan

REFERENCES:
- [Derived] Davies BR, Guan N, Logie A, Crafter C, Hanson L, Jacobs V, James N, Dudley P, Jacques K, Ladd B, D'Cruz CM, Zinda M, Lindemann J, Kodaira M, Tamura K, Jenkins EL. Tumors with AKT1E17K Mutations Are Rational Targets for Single Agent or Combination Therapy with AKT Inhibitors. Mol Cancer Ther. 2015 Nov;14(11):2441-51. doi: 10.1158/1535-7163.MCT-15-0230. Epub 2015 Sep 8. PMID 26351323
- See also: d3610c00004_protocol_protocol amendments_Redacted_JPOL MP 11APR_Redacted....pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1364&filename=d3610c00004_protocol_protocol%20amendments_Redacted_JPOL%20MP%2011APR_Redacted....pdf